CLINICAL TRIAL: NCT05225480
Title: Reinforcement of Placebo Response in Knee Osteoarthritis: A Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: Department of Psychology and Behavioural Sciences, Aarhus University (Unknown)
Responsible Party: Principal Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APPI2-OA-2022-01
Record Dates: First submitted 2022-01-13; First posted 2022-02-04 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
Keywords: Illness perception; Knee osteoarthritis; Placebo; Randomized trial
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: randomized single blind controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are masked as to which intervention (conversation) is considered the actual intervention. Therapists doing physical tests are blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): The illness perception conversation will be delivered in one session during around 15 minutes. The conversation will be based on responses to the eight item Brief illness perception questionnaire and a rating of the most relevant item made by the patient on the same day.
  The aim of the conversation will be to get an overview of the patient's illness perceptions concerning their knee OA and what is deemed the most maladaptive perceptions by the participant. Participants will be invited to elaborate on their thoughts concerning these perceptions.Although any maladaptive perceptions will be corrected if natural during the conversation, the conversation will not lead to any active attempts of changing illness perceptions. Rather, the conversation focusses on giving patients time and opportunity to express knee pain related perceptions and worries concerning their knee pain.
  Interventions: Behavioral: Illness perception conversation
- control arm (Active Comparator): The control conversation will be delivered in one session during around 15 minutes. In order to create two similar conversational settings where the only difference is the actual content of the conversations. The conversation will be based on responses to an eight item questionnaire concerning motivation for research participation and - similar to the illnes perception conversation - a rating of the most relevant item made by the patient.
  The aim of the conversation will be to get an overview of the patient's motivation for research participation and let them elaborate on their thoughts concerning their motivation.
  Interventions: Behavioral: research motivation conversation

INTERVENTIONS:
Behavioral: Illness perception conversation — A conversation based on the indvidual's knee pain related illness perceptions
  Arms: intervention arm
Behavioral: research motivation conversation — A conversation based on the indvidual's motivation for participating in research
  Arms: control arm

SUMMARY:
Saline intra-articular injections used as placebo treatments have been shown to provide pain relief in knee osteoarthritis (OA) It has further been shown that beneficial effects can be induced merely by having a conversation with a health professional.

The aim of this study is to determine whether an individual conversation based on the individual's illness perception related to knee OA affects the response to an intra-articular treatment with saline in individuals with knee OA.

DETAILED DESCRIPTION:
Despite many years of research, there is still considerable uncertainty on what causes placebo effects and how these are mediated. Saline is a pharmacologically inert agent frequently used as placebo comparator in clinical trials of intra-articular (IA) treatments for knee osteoarthritis (OA) and patients often experience a significant pain improvement from this treatment even when it is administered as an open label placebo treatment.

It has further been shown that beneficial effects can be induced merely by having a conversation with a health professional and several studies have found the alliance between therapist and patient to have a positive effect on treatment outcome in physical rehabilitation indicating that positive attention by itself leads to beneficial treatment outcomes. Still it is unclear wether the effect of an open label placebo treatment can be influenced by a conversation and if the extent of this infleuence depends on the focus of the conversation.

The aim of this study is to determine whether a conversation about the individual's illness perception related to knee OA affects the response to a placebo treatment (saline injection) in individuals with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* A clinical diagnosis of tibiofemoral OA in the target knee according to the American College of Rheumatology
* Average knee pain in the last week during weight bearing activities of at least 4 on a 0 to 10 points scale (0=no pain; 10=worst possible pain).

Exclusion Criteria:

* Not able to speak or understand Danish
* Scheduled surgery during study participation
* History of target knee surgery within 12 months
* History of arthroplasty in the target knee
* Injection therapy in either knee within 3 months
* Current use of oral glucocorticoids
* Current use of synthetic or non-synthetic opioids
* Contraindications to intra-articular injections, such as wounds or skin rash over injection site.
* Planning to start or discontinue other treatment for knee OA in the study participation period
* Inflammatory arthritis, such as rheumatoid arthritis or psoriatic arthritis.
* Regional pain syndromes
* Generalised pain syndromes such as fibromyalgia
* Lumbar or cervical nerve root compression syndromes
* Any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation, such as large knee joint effusion, uncontrolled diabetes, psychiatric and/or neurological disorders, or opiate dependency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
VAS knee pain | Week two, change from baseline
  Knee pain defined as "the average level of pain in your knee today" will be assessed with a 100 mm visual analogue scale (VAS) with anchors 0 = "no pain" and 100 = "Worst imaginable pain".

SECONDARY OUTCOMES:
The effect of knee pain variability (VAS) prior to the intervention | Week 0, Change from week -1
  The key secondary objective is to assess if pain variability in the week before treatment is a determinant of the effect of the subsequent treatment.
Brief Illness perception questionnaire | Week two, change from baseline
  The Brief illness perception questionnaire (BIPQ) is a generic questionnaire developed to measure illness perception in a variety of illnesses. The questionnaire is patient-reported and assesses perceptions on the following five dimensions: Identity, Cause, Timeline, Consequences and Cure-Control. It contains eight numerical rating scales questions (0-10) and a memo field based on the patients' own beliefs about their condition. In some circumstances it may be possible to compute an overall score which represents the degree to which the illness is perceived as threatening or benign. To compute the score, reverse score items 3, 4, and 7 and add these to items 1, 2, 5, 6, and 8. A higher score reflects a more threatening view of the illness.
Knee injury and Osteoarthritis Outcome Score | Week two, change from baseline
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is used to assess patient-reported knee-related symptoms. The KOOS is a patient-reported outcome measurement instrument developed to assess the patient's opinion about their knee and associated problems.KOOS comprises of 42 items in 5 separately scored subdomains: KOOS Pain (9 items), KOOS Symptoms (7 items), Function in daily living (KOOS Function; 17 items), Function in Sport and Recreation (5 items), and Knee-related Quality of Life (4 items). The previous week is the time period considered when answering the questions, and the questions relate to one knee (the target knee in this trial).
The 30 seconds sit to stand test | Week two, end of trial, change from baseline
  The 30 seconds chair stand test (30sCST) is a physical performance test that quantifies how many sit-to-stand movements an individual can perform within 30 seconds. The 30sCST is a measure of balance 500 during functional activities and lower extremity function and strength. It is recommended as a 501 performance-based test to assess physical function in people diagnosed with hip or knee OA. From the sitting position in the middle of seat with feet shoulder width apart, flat on the floor, arms crossed at chest, the participant is asked to stand completely up, then sit completely back down, repeatedly for 30 seconds. The total number of complete chair stands (up and down represents one stand) is counted. There is given only one trial. If a full stand is completed at 30 seconds, then this is counted in the total. The same chair is used at all assessments.
4x10 meter fast walk test | Week two, change from baseline
  The 4x10 meter fast walk test (40mFWT) is a physical performance test that quantifies short distance walking performance. The 40mFWT is a measure of walking speed over short distances and changing direction during walking. It is recommended as a performance-based test to assess physical function in people diagnosed with hip or knee OA (26).
  The participant is asked to walk as quickly but as safely as possible to a mark 10 m away, return, and repeat for a total distance of 40 m. Regular walking aid is allowed and recorded. Time of one trial, with turn time excluded, is recorded and expressed as speed m/s by dividing distance (40 m) by time (s).
Stair climbing test | Week two, change from baseline
  A stair climbing test (SCT) is a physical performance test that quantifies how fast an individual can ascend and descend a flight of stairs in a usual manner. The SCT is a measure of balance during functional activities and lower extremity function and strength. It is recommended as a performance-based test to assess physical function in people diagnosed with hip or knee OA.
  The participant is asked to ascend and descend a flight of stairs in a usual manner, and at a safe and comfortable pace. Use of any walking aid and handrail is permitted and recorded. Total time to ascend and descend steps for one trial is recorded in seconds. The same flight of stairs is used at all assessments.
Expectations for Treatment Scale (ETS) | Week 0, change from week -1
  The expectation for treatment scale (ETS) is a 5-item questionnaire concerning the patients' expectations of a given treatment. (E.g: 1) "I expect the treatment will help me to cope with my complaints", 2) "I expect the treatment will make my complaints disappear", 3) I expect the treatment will improve my energy", 4) "I expect the treatment will improve my physical performance" and 5) "I expect that after the treatment, my complaints will be considerably better".
  Each question has four response options on a likert scale: "partially disagree", "partially agree","agree", "definitely agree".
  We will replace the word "treatment" with "saline injection" and "complaint" with "knee pain". The questionnaire has been translated into Danish for this study.
Synovial hypertrophy score | Week two, change from baseline
  Via ultrasound, the amount of synovial hypertrophy will be measured in mm in position using specific landmarks. The following positions will be examined: 1) The medial joint space and recess (medial longitudinal scan) 2) The lateral joint space and recess (lateral longitudinal scan)
Doppler activity score | Week two, change from baseline
  Via ultrasound, the Doppler activity will be measured on a semi-quantitative score from 0-3.
Self-reported paracetamol and ibuprofen use for knee pain | Week two, change from baseline
  Participants will register their daily use of paracetamol and ibuprofen for knee pain

OTHER OUTCOMES:
Knee joint effusion | Week two, change from baseline
  As a safety outcome, the presence of knee joint effusion will be recorded for each knee as a dichotomous score (present/absent) using ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, Professor, Principal Investigator — the Parker Institute, Bisbebjerg and Frederiksberg Hospital
Locations (1):
- The Parker Institute, Bispebjerg-Frederiksberg Hospital, Frederiksberg, Danmark, Denmark

REFERENCES:
- [Derived] Ginnerup-Nielsen E, Jorgensen TS, Dew-Hattens C, Christensen R, Berg JI, Vase L, Dossing A, Nielsen SM, Kristensen LE, Bliddal H, Ellegaard K, Henriksen M. The impact of an illness perception conversation on open-label placebo response in knee osteoarthritis: A randomised controlled trial. Osteoarthritis Cartilage. 2024 Dec;32(12):1610-1619. doi: 10.1016/j.joca.2024.07.005. Epub 2024 Jul 17. PMID 39029733